CLINICAL TRIAL: NCT02806310
Title: Clinical Predictive Value of Podocan and Wnt Regulatory Molecules in Development of Aortopathy in Bicuspid Aortic Valve Disease
Brief Title: Podocan and Wnt Pathway in the Development of Aortopathy in Bicuspid Valve Disease
Status: Completed | Type: Observational
Sponsor: Bassett Healthcare (Other)
Responsible Party: Principal Investigator, Daniel Katz, Attending Physician - Cardiology, Bassett Healthcare
Other Study IDs: 2041
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Aortic Valve Disease
Keywords: Aortic Valve; Bicuspid
MeSH Terms: conditions — Aortic Valve Disease; Bicuspid Aortic Valve Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — All patients who do undergo valve replacement or aortic graft surgery within the 24 month follow up period, will have their valve tissue samples analyzed for podocan levels. These tissues are removed as a routine part of the surgery and sent to the clinical laboratory at Bassett. The Bassett Clinical Lab will prepare additional paraffin blocks and slides of the tissue for the research study. Specifically, aortic aneurysm and aortic root tissue will be analyzed. The relationship between cell density (mm2) and Podocan, in addition to the six Wnt molecule levels, will be analyzed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prospective: Group A: Patients with known BAV who are scheduled to have a cardiac MRI.
  Interventions: Other: Blood draw
- Historic: Group B: Patients with known BAV who have already had an MRI within the past year
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — blood sampling for biomarker levels

SUMMARY:
Bicuspid Aortic Valve (BAV) disease is a common cardiac anomaly that is associated with valvular abnormalities, both stenosis and regurgitation, and aortopathy. It is also shown to play role in abnormal aortic distensibility and stiffness with impairment of aortic elasticity and Left ventricular dysfunction. Mechanism of aortopathy is complex and is not understood completely. In a recent study podocan is found in extracellular matrix (ECM) of human aorta and is found to be accumulated in human abdominal aortic aneurysms. There is no current effective therapy that can alter the progression of aortic dilatation in bicuspid valve disease. Aortic surgery and aortoplasty is the only treatment in severely dilated aorta and aortic dissection. In this study the aim is to investigate the association between podocan and Wnt pathway in development and pathogenesis of aortopathy. This could provide more effective and physiological understanding of disease process and potential target in prevention and treatment for aortopathy.

DETAILED DESCRIPTION:
Patients with known BAV will be enrolled in two inclusion criteria categories:

- Group A: Patients who are scheduled to have a cardiac MRI

Procedures for Group A: MRI will be used as a standard procedure to confirm the morphology of bicuspid valve especially in uncertain cases and to do accurate aortic measurements. Patients who agree to participate will provide informed consent prior to their cardiac MRI/CT. A 6 minute walk test to measure baseline functional status will be performed after consent. All patients having a cardiac MRI/CT have an IV line placed as normal procedure. When then line has been placed, prior to contrast infusion a blood sample will be collected to test for circulatory Podocan and Wnt pathway molecules. At 24 months post procedure the following information will be collected from the participants' charts for endpoint analysis:

* All cause mortality
* Hospital admissions for Aortic dissection, Congestive heart failure, endocarditis or cardiac death
* Valve replacement or aortic graft surgery

  * Group B: Patients who have already had an MRI within the past year

Procedures for Group B: MRI will be used as a standard procedure to confirm the morphology of bicuspid valve especially in uncertain cases and to do accurate aortic measurements. Patients who agree to participate will report to the Clinical Research Division (CRD ) for a research visit to enroll in the study. At this visit, the patient will provide informed consent, complete a 6 minute walk test to measure baseline functional status , and will have blood drawn by venipuncture to obtain a blood sample to test for circulatory Podocan and Wnt pathway molecules. At 24 months post procedure the following information will be collected from the participants' charts for endpoint analysis:

* All cause mortality
* Hospital admissions for Aortic dissection, Congestive heart failure, endocarditis or cardiac death
* Valve replacement or aortic graft surgery

All patients who do undergo valve replacement or aortic graft surgery within the 24 month follow up period, will have their valve tissue samples analyzed for podocan levels. These tissues are removed as a routine part of the surgery and sent to the clinical laboratory at Bassett. The number of tissue samples collected during this procedure can range from one to four based on the exact nature and location of the aortic pathology. The Bassett Clinical Lab will prepare additional paraffin blocks and slides of the tissue for the research study.

A blood sample will also be taken at the time of the patient's post-op MRI to test for circulatory Podocan and Wnt pathway molecules. This usually occurs about 6-9 months after surgery.

It is expected that 100 participants will be enrolled in the study over 18 months. This is a sample size of convenience for this pilot study based the current volume of patients undergoing cardiac MRI/CT for evaluation of valvular disease. Of these 100 patients, it is estimated that 25 will undergo surgery as described above within the study period.

Baseline analysis will be performed to study the association between circulatory Podocan and Wnt regulatory molecules (Wnt-1, Wnt-3, Dkk-1, WIF-1, sFRP-1, sFRP-3) measured by ELISA in peripheral blood and tissue samples of aortic root/ascending aorta.

Each participant's chart will be reviewed at the time of enrollment and the following variables will be abstracted from the medical record:

* age,
* gender,
* ethnicity,
* Most recent Ht, Wt, BP, HR
* BMI
* Tobacco use/history
* Alcohol use/ history
* Comorbidities

  * HTN
  * Hyperlipidemia
  * Diabetes
  * CKD
  * Cancer
  * CAD
* Info from previous echocardiogram:

  * Ejection fraction
  * Valve area
  * Gradient
* Info from previous cardiac cath (if done):

  * Presence/absence of coronary stenosis
  * Location and degree of stenosis
  * Aortic valve area
  * Calculation of valve area
* Info from previous ECG:

  * Rhythm
  * LVH
* Medications
* Laboratory data:

  * Lipids
  * Chemistries
  * CBC
  * HgA1C
  * Troponin
  * BNP

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Patients with known BAV diagnosed by echocardiography, previous MRI, or cardiac CT
* Scheduled for cardiac MRI or have had a cardiac MRI within the past year
* Able to provide informed consent
* Ambulatory and expected to be able to complete 6 minute walk test

Exclusion Criteria:

* Patients without BAV
* Patients who have already had surgery for aortic valve problems and/or aortopathy
* Unable to complete 6 minute walk test (ex. Wheelchair bound)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known BAV.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Circulatory podocon levels | Day 1
circulatory WNT pathway molecule levels | Day1

SECONDARY OUTCOMES:
podocon expression in aortic tissue | 24 months
WNT pathway molecule expression in aortic tissue | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: daniel Katz, MD, Principal Investigator — Bassett Healthcare
Locations (1):
- Bassett Healthcare Network, Cooperstown, New York, United States

IPD SHARING:
Plan to Share IPD: No